CLINICAL TRIAL: NCT02778893
Title: A Phase Ⅳ,Open,Multicenter,Single Arm Study to Evaluate the Efficacy of the Combination Conmana With Thalidomide in Patients With NSCLC(Non-Small-Cell-Lung-Cancer)
Brief Title: Conmana Combined With Thalidomide to Treat NSCLC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, XiaoJu Zhang, Chief Physician, Henan Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: ICO-01
Record Dates: First submitted 2016-05-11; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: NSCLC
Keywords: Conmana; Thalidomide; NSCLC; EGFR mutation
MeSH Terms: interventions — icotinib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conmana and Thalidomide (Experimental): Conmana(Icotinib Hydrochloride Tablets) and Thalidomide:
  Conmana(Icotinib Hydrochloride Tablets) will be administered at 125mg three times a day(TID）continuously; Thalidomide will be administered at 100mg one a day（QD)at night continuously,If can tolerance after 1 weeks to add to 200mg.
  Interventions: Drug: Conmana; Drug: Thalidomide

INTERVENTIONS:
Drug: Conmana — 125mg three times a day (TID) continuously
  Other Names: Icotinib; Icotinib Hydrochloride Tablets
Drug: Thalidomide — 100mg one a day（QD）at night continuously,If can tolerance after 1 weeks to add to 200mg;
  Other Names: Sedoval; Thalomid; Celgene Brand of Thalidomide

SUMMARY:
Our study the NSCLC harbors EGFR-mutation with Conmana combined with thalidomide as first-line treatment, is expected to improve further EGFR-Tyrosine kinase inhibitors (TKI) response rate (ORR), prolong time to progression (PFS), improve patient survival.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy, survival and side effects of the combined therapy, and to evaluate the effectiveness and safety of thalidomide with Conmana in patients who harbors EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and the willingness to sign a written informed consent document.
2. Patients be age >18 years and < 75 years. Patients must have a Life Expectancy of greater than 3 months.
3. Patients must be NSCLC confirmed by Histological or cytological.
4. Eastern Cooperative Oncology Group (ECOG) score standard: 0-2.
5. Patients must have normal organ and marrow function as defined below, within two week prior to study: absolute neutrophil count>1,500/mL platelets>100,000/mL total bilirubin: within normal institutional limits Aspartate transaminase (AST)/Alanine aminotransferase (ALT) <2.5 times institutional upper limit of normal creatinine≤1.5 times institutional upper limit of normal urine dipstick for proteinuria of < less than 1+. If urine dipstick is > 1+ then a 24 hour urine for protein must demonstrate <500mg of protein in 24 hours to allow participation in the study.
6. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Judging by the researchers, that patients can comply with the program.

Exclusion Criteria:

1. Women that are pregnant or breastfeeding Note: Pregnant women are excluded from this study because the agents used in this study may be teratogenic to a fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with thalidomide, breastfeeding women are also excluded from this study.
2. During the course of the treatment, the serious active infection of intravenous injection of antibiotics is required.
3. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to thalidomide and icotinib or other agents used in the study are excluded.
4. A person who is not effectively controlled, has symptoms of brain metastases, or suffers from a mental disorder that is not easily controlled; has a severe mental or cognitive impairment.
5. Congestive heart failure, arrhythmia, myocardial infarction, unstable angina, stroke or transient ischemic attack in 6 months.
6. 5 years of suffering from other malignancies, except for the treatment of cervical carcinoma in situ or skin squamous cell carcinoma of the skin, or the basic control of skin basal cell carcinoma.
7. Can not follow the test program or can not meet the follow-up of patients.
8. The researchers think it is not appropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
5 years the progression-free survival (PFS) rate of the combination of thalidomide with gefitinib in patients who harbors EGFR mutations. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- XZhang, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes